CLINICAL TRIAL: NCT07218263
Title: Efficacy of a Novel Web-based Fatigue and Cognitive Assessment Platform in Detecting Fatigue and Depression
Brief Title: AI Platform for Fatigue and Depression Detection
Status: Not yet recruiting | Type: Observational
Sponsor: Brijesh Patel (Other)
Collaborators: SmartTec Inc (Industry)
Responsible Party: Sponsor-Investigator, Brijesh Patel, Assistant Professor of Clinical Medicine, Indiana University
Organization: Indiana University (Other)
Other Study IDs: IU-Okaya-2025; IRB #25854 (Other: Indiana University)
Record Dates: First submitted 2025-10-13; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Depression Disorders; Fatigue Symptom; Cardiovascular
Keywords: Fatigue; Depression; Artificial Intelligence
MeSH Terms: conditions — Fatigue; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Assignment: Participants will complete PHQ-9, FAS, and Okaya assessments.
  Interventions: Diagnostic Test: Participants will complete PHQ-9, FAS, and Okaya assessments.

INTERVENTIONS:
Diagnostic Test: Participants will complete PHQ-9, FAS, and Okaya assessments. — AI-based conversational assessment using facial and vocal features to evaluate fatigue and depression.

SUMMARY:
This observational study evaluates the accuracy of the Okaya AI platform in detecting fatigue and depression in cardiology patients, comparing its assessments to PHQ-9 and Fatigue Assessment Scale scores.

DETAILED DESCRIPTION:
Patients frequently experience fatigue and depression, which are often underdiagnosed due to limitations in traditional screening tools. This study introduces the Okaya platform, a browser-based AI system that analyzes facial and vocal biomarkers collected during conversational check-ins. The platform uses computer vision and natural language processing to extract features such as eye contact, facial affect, pitch, volume, and speech patterns. These features are processed through regression models to generate a composite AI based score. The study aims to validate this score against PHQ-9 and FAS assessments. Participants will complete a single baseline check-in using the Okaya platform and complete standard questionnaires. No interventions will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18, English-speaking, able to consent

Exclusion Criteria:

* Active substance use, nonverbal, cognitive disability, active suicidal/homicidal ideation

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants will be selected from both inpatient and outpatient setting.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Correlation between Okaya (AI based) score and PHQ-9 | Baseline
  Regression analysis comparing Okaya scores to PHQ-9
Correlation between Okaya (AI) based score and PHQ-9 and FAS | Baseline
  Regression analysis comparing Okaya scores to standard assessments
Correlation between Okaya (AI based) score and FAS | Baseline
  Regression analysis comparing Okaya scores to FAS

SECONDARY OUTCOMES:
Usability and patient satisfaction | Baseline
  Ease-of-use ratings on the Okaya platform

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No